CLINICAL TRIAL: NCT00584441
Title: Menstrual Differences in Airway Inflammation in Asthma
Status: Completed | Type: Observational
Sponsor: The University of Texas Medical Branch, Galveston (Other)
Responsible Party: Sponsor
Other Study IDs: 07-256
Record Dates: First submitted 2007-12-20; First posted 2008-01-02 (Estimated); Last update posted 2013-02-13 (Estimated); Status verified 2013-02

CONDITIONS: Asthma
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Serum Eosinophil Cationic Protein (ECP) samples will be obtained. The 5ml blood samples for measuring ECP levels will be collected in silica gel-containing tubes. After centrifuging, the supernatant will be frozen and ECP levels will bemeasured using an ELISA kit
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- 1: Women with pre-menstrual asthma (PMA): As defined by a 20% or more fall in PEFR and / or change by 20% or more of daily symptom score.
- 2: Women without pre-menstrual asthma
- 3: Women on oral contraceptives

SUMMARY:
Asthma is a chronic inflammatory lung disease characterized by airway hyper-responsiveness and reversible airway obstruction. Over the last decade, the prevalence of asthma is on the rise and it disproportionately affects more women than men. As much as 40% of women with asthma are known to have worsening of asthma symptoms and lung function prior to menstruation. This syndrome is being increasingly recognized as premenstrual asthma (PMA). The pathologic differences in female asthmatics with and without this syndrome are not known. The evidence regarding the role of sex hormones has been contradicting. We propose an observational cohort study to examine the changes in airway inflammation in women with asthma in relation to their menstrual cycle and their association with sex hormone levels. In addition we will include women on oral contraceptives to determine their effect on airway inflammation and asthma symptoms.

We hypothesis that:

* Women with premenstrual asthma will show increased indices of airway inflammation in various phases the monthly menstrual cycle.
* In women with premenstrual asthma, a change in serum estradiol/progesterone ratio during the late luteal phase is associated with worsening of airway inflammation, air flow limitation and asthma symptoms.
* The use of oral contraceptives is associated with suppression of the cyclical changes in airway inflammation due to lack of fluctuations in estradiol and progesterone levels.

Recruited subjects will be asked to record asthma symptom scores, morning Peak Expiratory Flow Rate (m-PEFR) and rescue asthma medication (β2-agonist) used daily during the one month screening period to identify women with and without pre-menstrual asthma. Asthmatic women with regular menstrual cycles will be evaluated in their follicular phase (days 5-8) and luteal phase (days 21-24) and women on oral contraceptive pills (OCP) will be evaluated on days 9-12 of their OCP cycle and during the days 25-28, off of OCP consecutively for a 2-month period.

ELIGIBILITY:
Inclusion Criteria:

* With diagnosis of Asthma (ICD-9 Code 493)
* Requiring low to moderate dose inhaled corticosteroids for control.
* With Pre-bronchodilator FEV1 ≥50% and ≤90% of predicted normal
* With a positive bronchodilator response
* Non smoker or Ex-smoker (Quit >1 year ago)
* Regular menstrual cycle (24-35 days cycle)
* With and without OCP use
* Constant dose of asthma maintenance medication for at least 30 days prior to enrolment

Exclusion Criteria:

* Recent use of systemic steroids (<30 days)
* Severe Asthma (FEV1 <50% or frequent exacerbations or systemic steroid dependence)
* Negative bronchodilator response
* Current Smoker
* Irregular Menses or postmenopausal
* Positive pregnancy test
* Use of hormonal contraceptives other than monophasic OCPs
* Exacerbation or Respiratory Infection or antibiotic use within the last 30 days

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Females diagnosed with asthma, with either regular menstral cycles or on monophasic oral contraceptives, with or without pre-mentstual asthma symptoms
Sampling Method: Non-Probability Sample
Enrollment: 6 (Actual)
Dates: Start 2007-09; Primary Completion 2010-02 (Actual); Study Completion 2010-02 (Actual)

PRIMARY OUTCOMES:
To evaluate menstrual-related changes in airway inflammation of asthma patients with and without premenstrual worsening of symptoms. | 3 months

SECONDARY OUTCOMES:
To examine the effect of sex hormones in airway inflammation | 3 months
To examine the effect of oral contraceptive pills on airway inflammation | 3 months
To assess the cyclical changes in airway inflammation as measured by -Fractional exhaled Nitric Oxide (FeNO), -Exhaled Breath Condensate (EBC) pH and -Serum eosinophil cationic protein (ECP), in asthmatic women with and without premenstrual asthma. | 3 months
To analyze the association of between serum estradiol and progesterone levels and the variation in airway inflammation, airflow limitation and asthma symptoms | 3 months
To study the effect of oral contraceptives on airway inflammation by measuring serum and exhaled inflammatory indices | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Anandhi T Murugan, MD, MPH, Principal Investigator — University of Texas
Locations (1):
- University of Texas Medical Branch, Galveston, Texas, United States